CLINICAL TRIAL: NCT00166101
Title: Near Infrared Spectroscopy Monitoring of Cerebral Oxygen Saturation in Neonatal Cardiac Surgery - Comparison With Common Methods of Estimating Adequate Systemic Perfusion
Brief Title: NIRS in Neonatal Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Steven R Tosone MD, Assistant Professor, Emory University
Other Study IDs: 459-2002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Hypoplastic Left Heart; Surgery
Keywords: pediatric; cardiac surgery
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to the small size of infants and the use of bypass machines, physicians have difficulty assessing whether the infant's brain and body is getting enough oxygen during heart surgery. This study compares continuous monitoring via the NIRS (Near Infrared Spectroscopy) to the traditional methods of determining oxygen saturation.

DETAILED DESCRIPTION:
One of the limiting factors in treating infants undergoing cardiac surgery is the difficulty in assessing systemic perfusion with accuracy. At Children's Healthcare of Atlanta, Near-infrared Spectroscopy (NIRS) is available, but has never been studied. In patients undergoing first stage palliation (Norwood) for hypoplastic left heart, routine management will be utilized in addition to the NIRS monitor. The following will be documented pre- and post-bypass, then every 4 hours for 24 hours after admission to the Cardiac Intensive Care Unit:NIRS readings, Lactic acid levels,mixed venous saturations,hemoglobin, hematocrit, arterial blood gases, heart rate, blood pressure, central venous pressure, left atrium pressure,core temperature, toe temperature, pulse oximeter reading, urine output, ventilator settings, inotropic levels. All the data will be entered into a database and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* hypoplastic left heart
* requiring stage 1 palliation
* informed consent obtained

Exclusion Criteria:

* does not have hypoplastic left heart
* is not having stage 1 palliation
* no informed consent

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with Hypoplastic Left Heart Syndrome undergoing stage 1 palliation with the Norwood procedure.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2002-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Tosone, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Adcock LM, Wafelman LS, Hegemier S, Moise AA, Speer ME, Contant CF, Goddard-Finegold J. Neonatal intensive care applications of near-infrared spectroscopy. Clin Perinatol. 1999 Dec;26(4):893-903, ix. PMID 10572728
- [Background] Madsen PL, Secher NH. Near-infrared oximetry of the brain. Prog Neurobiol. 1999 Aug;58(6):541-60. doi: 10.1016/s0301-0082(98)00093-8. PMID 10408656
- [Background] Kurth CD, Steven JM, Nicolson SC. Cerebral oxygenation during pediatric cardiac surgery using deep hypothermic circulatory arrest. Anesthesiology. 1995 Jan;82(1):74-82. doi: 10.1097/00000542-199501000-00011. PMID 7832338
- [Background] Nollert G, Shin'oka T, Nagashima M, Shum-Tim D. Cerebral oxygenation during cardiopulmonary bypass in children. J Thorac Cardiovasc Surg. 1997 Nov;114(5):871-3. doi: 10.1016/S0022-5223(97)70105-3. No abstract available. PMID 9375629
- [Background] Daubeney PE, Pilkington SN, Janke E, Charlton GA, Smith DC, Webber SA. Cerebral oxygenation measured by near-infrared spectroscopy: comparison with jugular bulb oximetry. Ann Thorac Surg. 1996 Mar;61(3):930-4. doi: 10.1016/0003-4975(95)01186-2. PMID 8619720
- [Background] Wardle SP, Yoxall CW, Weindling AM. Determinants of cerebral fractional oxygen extraction using near infrared spectroscopy in preterm neonates. J Cereb Blood Flow Metab. 2000 Feb;20(2):272-9. doi: 10.1097/00004647-200002000-00008. PMID 10698064
- [Background] Daubeney PE, Smith DC, Pilkington SN, Lamb RK, Monro JL, Tsang VT, Livesey SA, Webber SA. Cerebral oxygenation during paediatric cardiac surgery: identification of vulnerable periods using near infrared spectroscopy. Eur J Cardiothorac Surg. 1998 Apr;13(4):370-7. doi: 10.1016/s1010-7940(98)00024-4. PMID 9641334
- [Background] Kurth CD, Steven JM, Nicolson SC, Chance B, Delivoria-Papadopoulos M. Kinetics of cerebral deoxygenation during deep hypothermic circulatory arrest in neonates. Anesthesiology. 1992 Oct;77(4):656-61. doi: 10.1097/00000542-199210000-00007. PMID 1416162
- [Background] Watzman HM, Kurth CD, Montenegro LM, Rome J, Steven JM, Nicolson SC. Arterial and venous contributions to near-infrared cerebral oximetry. Anesthesiology. 2000 Oct;93(4):947-53. doi: 10.1097/00000542-200010000-00012. PMID 11020744
- [Background] du Plessis AJ, Newburger J, Jonas RA, Hickey P, Naruse H, Tsuji M, Walsh A, Walter G, Wypij D, Volpe JJ. Cerebral oxygen supply and utilization during infant cardiac surgery. Ann Neurol. 1995 Apr;37(4):488-97. doi: 10.1002/ana.410370411. PMID 7717685